CLINICAL TRIAL: NCT06735664
Title: A Phase I Study of Covalent BTK Inhibitor Zanubrutinib in Combination With a CD3-CD20 Bispecific Antibody Odronextamab in Patients With Richter's Transformation
Brief Title: Zanubrutinib in Combination With Odronextamab for the Treatment of Patients With Richter's Transformation
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 23667; NCI-2024-10074 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 23667 (Other: City of Hope Medical Center); P30CA033572 (NIH)
Record Dates: First submitted 2024-12-11; First posted 2024-12-16 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Recurrent Transformed Chronic Lymphocytic Leukemia; Refractory Transformed Chronic Lymphocytic Leukemia; Richter Syndrome; Transformed Chronic Lymphocytic Leukemia to Diffuse Large B-Cell Lymphoma
MeSH Terms: interventions — Biopsy; Specimen Handling; Magnetic Resonance Spectroscopy; High-Energy Shock Waves; zanubrutinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (odronextamab, zanubrutinib) (Experimental): Patients receive odronextamab IV over 4 hours on days 1, 2, 8, 9, 15 and 16 of cycle 1 and over 1-4 hours on days 1, 8 and 15 of cycles 2-4 and then on days 1 and 15 of remaining cycles. Patients with CR at cycle 9 may receive odronextamab on day 1 of remaining cycles. Starting with cycle 2, patients also receive zanubrutinib PO QD or BID of each cycle. Cycles repeat every 21 days for cycles 1-4 in the absence of disease progression or unacceptable toxicity then repeat every 28 days for up to cycle 12. After 12 cycles, patients may continue zanubrutinib at investigator's discretion. Patients also undergo ECHO or MUGA and optional bone marrow biopsy at screening and ultrasound guided biopsy of lymph node at screening and during days 2-12 of cycle 2. Additionally, patients undergo blood sample collection and PET, or CT throughout the study.
  Interventions: Procedure: Biopsy; Procedure: Biospecimen Collection; Procedure: Bone Marrow Biopsy; Procedure: Computed Tomography; Procedure: Echocardiography; Procedure: Multigated Acquisition Scan; Biological: Odronextamab; Procedure: Positron Emission Tomography; Procedure: Ultrasound Imaging; Drug: Zanubrutinib

INTERVENTIONS:
Procedure: Biopsy — Undergo ultrasound guided biopsy
  Other Names: BIOPSY_TYPE; Bx
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Bone Marrow Biopsy — Undergo optional bone marrow biopsy
  Other Names: Biopsy of Bone Marrow; Biopsy, Bone Marrow
Procedure: Computed Tomography — Undergo CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; tomography
Procedure: Echocardiography — Undergo ECHO
  Other Names: EC
Procedure: Multigated Acquisition Scan — Undergo MUGA
  Other Names: Blood Pool Scan; Equilibrium Radionuclide Angiography; Gated Blood Pool Imaging; Gated Heart Pool Scan; MUGA; MUGA Scan; Multi-Gated Acquisition Scan; Radionuclide Ventriculogram Scan; Radionuclide Ventriculography; RNV Scan; RNVG; SYMA Scanning; Synchronized Multigated Acquisition Scanning
Biological: Odronextamab — Given IV
  Other Names: Anti-CD20 x Anti-CD3 Bispecific Monoclonal Antibody REGN1979; REGN1979; WHO 11035
Procedure: Positron Emission Tomography — Undergo PET
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET Scan; Positron emission tomography (procedure); Positron Emission Tomography Scan; Positron-Emission Tomography; proton magnetic resonance spectroscopic imaging; PT
Procedure: Ultrasound Imaging — Undergo ultrasound guided biopsy
  Other Names: 2-Dimensional Grayscale Ultrasound Imaging; 2-Dimensional Ultrasound Imaging; 2D-US; Ultrasonography; Ultrasound; Ultrasound Test; Ultrasound, Medical; US
Drug: Zanubrutinib — Given PO
  Other Names: BGB 3111; BGB-3111; BGB3111; Brukinsa; BTK-InhB

SUMMARY:
This phase I trial tests the safety and side effects of zanubrutinib in combination with odronextamab and how well it works in treating patients with Richter's transformation. Zanubrutinib, a tyrosine kinase inhibitor, blocks a protein called Bruton tyrosine kinase (BTK), which may help keep cancer cells from growing. Odronextamab is a bispecific monoclonal antibody that can bind to two different antigens at the same time. Odronextamab binds to CD20 found on B-cells (a type of white blood cell) and on many B-cell cancers and to CD3 on T-cells (also a type of white blood cell) and may interfere with the ability of cancer cells to grow and spread. Giving zanubrutinib in combination with odronextamab may be safe, tolerable and/or effective in treating patients with Richter's transformation.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To evaluate safety and tolerability of zanubrutinib administered in combination with odronextamab in patients with Richter's transformation (RT).

SECONDARY OBJECTIVE:

I. To evaluate efficacy of zanubrutinib administered in combination with odronextamab, based on overall response rate (ORR), complete response (CR) rate, duration of response (DOR), progression-free survival (PFS), and overall survival (OS).

EXPLORATORY OBJECTIVE:

I. To characterize the T-cell population balance in patients treated with zanubrutinib and odronextamab.

OUTLINE:

Patients receive odronextamab intravenously (IV) over 4 hours on days 1, 2, 8, 9, 15 and 16 of cycle 1 and over 1-4 hours on days 1, 8 and 15 of cycles 2-4 and then on days 1 and 15 of remaining cycles. Patients with CR at cycle 9 may receive odronextamab on day 1 of remaining cycles. Starting with cycle 2, patients also receive zanubrutinib orally (PO) once daily (QD) or twice daily (BID) of each cycle. Cycles repeat every 21 days for cycles 1-4 in the absence of disease progression or unacceptable toxicity then repeat every 28 days for up to cycle 12. After 12 cycles, patients may continue zanubrutinib at investigator's discretion. Patients also undergo echocardiography (ECHO) or multigated acquisition scan (MUGA) and optional bone marrow biopsy at screening and ultrasound guided biopsy of lymph node at screening and during days 2-12 of cycle 2. Additionally, patients undergo blood sample collection and positron emission tomography (PET), or computed tomography (CT) throughout the study.

After completion of study treatment, patients are followed up at 4 and 12 weeks then every 6 months for up to 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Documented informed consent of the participant and/or legally authorized representative

  * Assent, when appropriate, will be obtained per institutional guidelines
* Age: ≥ 18 years
* Eastern Cooperative Oncology Group (ECOG) ≤ 2
* Histologically confirmed diagnosis of Richter transformation (RT; transformed CLL). Only patients who have diffuse large B-cell lymphoma histology in transformation are eligible (for example, patients with transformation into Hodgkin lymphoma subtype are not eligible)
* Evidence of CD20 positivity at screening (by immunohistochemistry [IHC] or flow cytometry)
* Treatment naïve or relapsed/ refractory disease. Patients with either previously untreated RT and previously treated RT are eligible, regardless of whether or not they had received CLL-directed therapy
* Radiographically measurable lymphadenopathy (≥ 1.5 cm) or splenomegaly, or bone marrow involvement by diffuse large B cell lymphoma (DLBCL)/RT
* Fully recovered from the acute toxic effects (except alopecia) to ≤ grade 1 to prior anti-cancer therapy
* Without bone marrow involvement: Absolute neutrophil count (ANC) ≥ 1,000/mm^3

  * NOTE: A participant may not have received granulocyte colony stimulating factor (G-CSF) within 3 days of first dose of the assigned study treatment in order to meet this eligibility requirement
* With bone marrow involvement: ANC ≥ 500/mm^3

  * NOTE: A participant may not have received granulocyte colony stimulating factor (G-CSF) within 3 days of first dose of the assigned study treatment in order to meet this eligibility requirement
* Without bone marrow involvement: Platelets ≥ 50,000/mm^3

  * NOTE: A participant may not have received platelet transfusion within 7 days of first dose of the assigned study treatment in order to meet this eligibility requirements
* With bone marrow involvement: Platelets ≥ 25,000/mm^3

  * NOTE: A participant may not have received platelet transfusion within 7 days of first dose of the assigned study treatment in order to meet this eligibility requirements
* With bone marrow involvement: Hemoglobin (Hgb) ≥ 7 g/dL
* Total bilirubin ≤ 2 x upper limit of normal (ULN) or ≤ 3 x ULN for Gilbert's disease or compensated hemolysis directly attributable to CLL
* Aspartate aminotransferase (AST) ≤ 3 x ULN
* Alanine aminotransferase (ALT) ≤ 3 x ULN
* Alkaline phosphatase (ALP) ≤ 2.5 x ULN or ≤ 5 x ULN if attributed to lymphoma involvement of the liver
* Serum creatinine ≤ 1.5 x ULN OR creatinine clearance of ≥ 50 mL/min per 24 hour urine test or the Cockcroft-Gault formula
* If not receiving anticoagulants: International normalized ratio (INR) OR prothrombin (PT) ≤ 1.5 x ULN
* If on anticoagulant therapy: PT must be within therapeutic range of intended use of anticoagulants
* If not receiving anticoagulants: Activated partial thromboplastin time (aPTT) ≤ 1.5 x ULN
* If on anticoagulant therapy: aPTT must be within therapeutic range of intended use of anticoagulants
* Left ventricular ejection fraction (LVEF) ≥ 45%

  * Note: To be performed within 28 days prior to day 1 of protocol therapy
* Seronegative for hepatitis C virus (HCV), hepatitis B virus (HBV) (surface antigen negative) and no history of HIV OR

  * If seropositive for HBV or HCV, nucleic acid quantitation must be performed. Viral load must be undetectable
  * HIV-infected patients on effective anti-retroviral therapy with undetectable viral load within 6 months are eligible for this trial
* Women of childbearing potential (WOCBP): Negative serum pregnancy test
* Agreement by females and males of childbearing potential to use an effective method of birth control or abstain from heterosexual activity for the course of the study through at least 6 months after the last dose of study therapy. Sperm donation is prohibited during the study and for 6 months after the last dose of the assigned study treatment. Highly effective contraceptive measures include:

  * Stable use of combined (estrogen and progestogen containing) hormonal contraception (oral, intravaginal, transdermal) or progestogen-only hormonal contraception (oral, injectable, implantable) associated with inhibition of ovulation initiated ≥ 2 menstrual cycles prior to screening
  * Intrauterine device (IUD); intrauterine hormone-releasing system (IUS)
  * Bilateral tubal ligation/occlusion
  * Vasectomized partner (provided that the male vasectomized partner is the sole sexual partner of the study patient and that the partner has obtained medical assessment of surgical success for the procedure)
  * Sexual abstinence, only if defined as refraining from heterosexual intercourse during the entire period of risk associated with the study drugs
  * Childbearing potential defined as not being surgically sterilized (men and women) or have not been free from menses for > 1 year (women only)
  * A postmenopausal state is defined as no menses for 12 months without an alternative medical cause. A high follicle stimulating hormone (FSH) level in the postmenopausal range may be used to confirm a postmenopausal state in women not using hormonal contraception or hormonal replacement therapy. However, in the absence of 12 months of amenorrhea, a single FSH measurement is insufficient to determine the occurrence of a postmenopausal state. The above definitions are according to the clinical trial facilitation group guidance. Pregnancy testing and contraception are not required

Exclusion Criteria:

* Allogeneic bone marrow or organ transplant within 6 months or evidence of active graft versus host diseae (GVHD)
* Prior CD20-targeted bispecific antibody therapy
* Chronic systemic corticosteroid use > 10 mg/day of prednisone or equivalent within 72 hours (h) of start of study treatment. Patients who received corticosteroid treatment with ≤ 10 mg/day of prednisone or equivalent must be documented to be on a stable dose of at least 4 weeks' duration prior to day 1 of cycle 1. Patients may have received a brief (≤ 10 days) course of systemic steroids (≤ 80 mg prednisone equivalent per day) up to 24 hours prior to initiation of study therapy for control of lymphoma-related symptoms
* Therapeutic anticancer antibodies within 2 weeks prior to day 1 of protocol therapy
* Radio- or toxin-immunoconjugates within 10 weeks prior to day 1 of protocol therapy
* Live vaccine within 28 days prior to day 1 of protocol therapy
* Any investigational therapy within 28 days or 5 half-lives of the drug, whichever is shorter, prior to the start of study treatment
* Standard radiotherapy within 14 days of first administration of study treatment
* Prior organ transplantation
* Chemotherapy, within 2 weeks prior to day 1 of protocol therapy; targeted therapy within 6 half-lives or two weeks, whichever is shorter
* Requires treatment with a strong CYP3A4 inducers/ inhibitor while on protocol therapy
* Uncontrolled immune hemolysis or thrombocytopenia
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to study drug
* Known hypersensitivity to both allopurinol and rasburicase
* Unstable cardiac disease as defined by one of the following:

  * Cardiac events such as myocardial infarction (MI) within the past 6 months
  * NYHA (New York Heart Association) heart failure class III-IV
  * Uncontrolled atrial fibrillation or hypertension
* Arterial or venous thrombotic or embolic events such as cerebrovascular accident (including transient ischemic attacks), deep vein thrombosis or pulmonary embolism within 3 months before the start of study treatment
* Unstable angina (angina symptoms at rest), new-onset angina (begun within the last 3 months)
* Active uncontrolled cardiac arrythmia
* History or concurrent condition of interstitial lung disease and/or severely impaired lung function
* Evidence of central nervous system (CNS) involvement within 6 months prior to initiation of study therapy
* Major surgery (under general anesthesia) within 30 days prior to day 1 of protocol therapy
* Clinically significant uncontrolled illness
* Evidence of any active infection (bacterial, viral, fungal, mycobacterial, parasitic or other) at study enrollment or within 2 weeks of study enrollment, if requiring ongoing treatment and/or has the potential to cause disseminated disease or severe infection upon immunosuppression. There should be evidence that the infection has cleared or is well controlled by start of study therapy
* Active COVID-19 infection
* Uncontrolled infection with human immunodeficiency virus (HIV), hepatitis B virus (HBV), or hepatitis C virus (HCV)

  * NOTE: Participants with HIV who have controlled infection (undetectable viral load and CD4 count above 350 cells/uL either spontaneously or on a stable antiviral regimen) are permitted
  * NOTE: Participants who are hepatitis B surface antigen positive or who are hepatitis B core antibody positive should undergo evaluation by a specialist and be considered to have controlled infection (serum hepatitis B virus deoxyribonucleic acid [DNA] polymerase chain reaction [PCR] that is below the limit of detection AND receiving anti-viral therapy for hepatitis B) before they are permitted onto study
  * NOTE: Participants who are HCV antibody positive who have controlled infection (undetectable HCV ribonucleic acid [RNA] by PCR either spontaneously or in response to a successful prior course of anti-HCV therapy) are permitted
* Cytomegalovirus (CMV) infection as noted by detectable levels on peripheral blood polymerase chain reaction (PCR) assay. Patients who show detectable levels of CMV at screening will need to be treated with appropriate antiviral therapy and demonstrate at least 2 undetectable levels of CMV by PCR assay (at least 7 days apart) before being re-considered for eligibility
* Other active malignancy. Patients with a prior (in the past 5 years) or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial. History of the following is allowed:

  * Malignancy treated with curative intent and no known active disease present for ≥ 2 years prior to initiation of therapy on current study
  * Adequately treated non-melanoma skin cancer or lentigo maligna (melanoma in situ) without evidence of disease
  * Adequately treated in situ carcinomas (e.g., cervical, esophageal, etc.) without evidence of disease
  * Asymptomatic prostate cancer managed with "watch and wait" strategy
* Females only: Pregnant or breastfeeding
* Inability to swallow and retain oral medication
* Any other condition that would, in the investigator's judgment, contraindicate the patient's participation in the clinical study due to safety concerns with clinical study procedures
* Prospective participants who, in the opinion of the investigator, may not be able to comply with all study procedures (including compliance issues related to feasibility/logistics)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Estimated)
Dates: Start 2025-08-14 (Actual); Primary Completion 2027-12-13 (Estimated); Study Completion 2027-12-13 (Estimated)

PRIMARY OUTCOMES:
Dose limiting toxicity (DLT) | During the first 2 cycles of protocol therapy (cycle length = 21 days)
  All non-hematologic toxicities will be coded and graded according to the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version (v) 5.0. Hematologic toxicities will be assessed per International Workshop on Chronic Lymphocytic Leukemia (IWCLL) 2018. Cytokine release syndrome (CRS)/immune effector cell associated neurotoxicity syndrome (ICANS) will be coded by American Society for Transplantation and Cellular Therapy (ASTCT) grading for CRS/ICANS. DLTs will be summarized by type, severity, and attribution. DLTs will be individually described.
Incidence of adverse events (AEs) | Up to 28 days after last dose of study treatment
  All non-hematologic toxicities will be coded and graded according to the NCI CTCAE v 5.0. Hematologic toxicities will be assessed per IWCLL 2018. CRS/ICANS will be coded by ASTCT grading for CRS/ICANS. AEs will be summarized by type, severity, and attribution.

SECONDARY OUTCOMES:
Overall response rate (ORR) | Up to 3 years
  ORR will be defined as the proportion of response evaluable patients who achieve a best response of complete response (CR) or partial response (PR) according to Lugano 2014 guidelines on study before any documented disease progression or any subsequent non-Hodgkin lymphoma (NHL) treatment. ORR will be estimated by the binary proportion, along with the 95% exact binomial confidence intervals (CIs).
CR rate | Up to 3 years
  Will be defined as the proportion of response evaluable patients who achieve a best response of complete response according to Lugano 2014 guidelines on study before any documented disease progression or any subsequent NHL treatment. CR rate will be estimated by the binary proportion, along with the 95% exact binomial CIs.
Duration of response (DOR) | From the first achievement of CR or PR to disease progression/relapse or death due to any cause, whichever is earlier, assessed up to 3 years
  Will be estimated using the product-limit method of Kaplan and Meier along with the Greenwood estimator of standard error; 95% CI will be constructed based on log-log transformation. Median DOR will be estimated when available.
Progression-free survival (PFS) | From start of protocol treatment to disease relapse/progression or death due to any cause, whichever is earlier, assessed up to 3 years
  Will be estimated using the product-limit method of Kaplan and Meier along with the Greenwood estimator of standard error; 95% CI will be constructed based on log-log transformation. Median PFS will be estimated when available.
Overall survival (OS) | From start of protocol treatment to death due to any cause, assessed up to 3 years
  Will be estimated using the product-limit method of Kaplan and Meier along with the Greenwood estimator of standard error; 95% CI will be constructed based on log-log transformation. Median OS will be estimated when available.

CONTACTS AND LOCATIONS:
Overall Officials: Alexey V Danilov, Principal Investigator — City of Hope Medical Center
Locations (1):
- City of Hope Medical Center, Duarte, California, United States